CLINICAL TRIAL: NCT05392621
Title: Optimizing Stress Management in College Students
Brief Title: Stress Management in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Jason Fanning, Assistant Professor, Wake Forest University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024664
Record Dates: First submitted 2022-05-13; First posted 2022-05-26 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Stress
Keywords: yoga; deep breathing; progressive muscle relaxation
MeSH Terms: interventions — Yoga; Autogenic Training

STUDY DESIGN:
Intervention Model Description: This is a 2x2x2 randomized factorial pilot trial. Participants will be randomized to receive one of 8 possible combinations of yoga (yes/no), progressive muscle relaxation (yes/no), or deep breathing (yes/no).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Yoga+Progressive Muscle Relaxation+Deep Breathing (Experimental): Participants engage in a single session combining yoga, progressive muscle relaxation, and deep breathing.
  Interventions: Behavioral: Yoga; Behavioral: Deep Breathing; Behavioral: Progressive Muscle Relaxation
- Yoga+Progressive Muscle Relaxation (Experimental): Participants engage in a single session combining yoga and progressive muscle relaxation
  Interventions: Behavioral: Yoga; Behavioral: Progressive Muscle Relaxation
- Yoga+Deep Breathing (Experimental): Participants engage in a single session combining yoga and deep breathing.
  Interventions: Behavioral: Yoga; Behavioral: Deep Breathing
- Yoga (Experimental): Participants engage in a single session of yoga.
  Interventions: Behavioral: Yoga
- Progressive Muscle Relaxation+Deep Breathing (Experimental): Participants engage in a single session combining progressive muscle relaxation and deep breathing.
  Interventions: Behavioral: Deep Breathing; Behavioral: Progressive Muscle Relaxation
- Progressive Muscle Relaxation (Experimental): Participants engage in a single session of progressive muscle relaxation.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Deep Breathing (Experimental): Participants engage in a single session of deep breathing.
  Interventions: Behavioral: Deep Breathing
- Quiet sitting (Sham Comparator): Participants engage in a low-touch relaxation condition.
  Interventions: Behavioral: Quiet sitting

INTERVENTIONS:
Behavioral: Yoga — A single Hatha yoga session designed to support stress management.
  Arms: Yoga; Yoga+Deep Breathing; Yoga+Progressive Muscle Relaxation; Yoga+Progressive Muscle Relaxation+Deep Breathing
Behavioral: Deep Breathing — A single deep breathing exercise session designed to elicit relaxation and to assist in stress management.
  Arms: Deep Breathing; Progressive Muscle Relaxation+Deep Breathing; Yoga+Deep Breathing; Yoga+Progressive Muscle Relaxation+Deep Breathing
Behavioral: Progressive Muscle Relaxation — A single session of progressive muscle relaxation designed to elicit relaxation.
  Arms: Progressive Muscle Relaxation; Progressive Muscle Relaxation+Deep Breathing; Yoga+Progressive Muscle Relaxation; Yoga+Progressive Muscle Relaxation+Deep Breathing
Behavioral: Quiet sitting — A single session of quiet sitting.
  Arms: Quiet sitting

SUMMARY:
Stress is defined as a response to one's evaluation of physical, emotional, or environmental challenges or demands. While the experience of stress is common, chronic exposure to high levels of stress is associated with a host of negative interrelated psychological, physiological, and behavioral outcomes. Mental health problems such as anxiety and depression have a high correlation with stress. In addition, chronic diseases such as cardiovascular disease are also thought to be related to stress. For instance, research shows that stress increases blood lipids by changing cholesterol levels eventually leading to arterial thrombosis and stroke.

While stress affects individuals across their lifespan, college students face a unique combination of academic and life challenges that exacerbate their experience of stress, making them highly susceptible to high levels of stress. Additionally, technological advances such as social media can be a source of chronic stress for many. As exposure to high levels of persistent stress is likely to predispose young adults to a lifetime of poor health and unhealthy behaviors, this is especially imperative in finding low impact and attainable methods of stress management for this population.

Although a significant body of literature has addressed stress reduction techniques, most studies to date focus on intervention effects that accumulate over months of exposure, with many stress management programs lasting at minimum of 8 weeks. Previous research has found that interventions employing yoga, progressive muscle relaxation (PMR), and deep breathing exercise (DBE) significantly reduce stress levels. The relationship between yoga and stress reduction has been especially consistent across studies. It has been suggested that mindfulness may be the active agent in such programs. Intriguingly, Fountain et al., (2019) found a single 20-minute yoga session significantly decreased stress levels in college students. This raises the question of whether yoga, PMR, and/or DBE require repeated exposure to provide helpful stress-reducing effects, or whether benefits may be obtained in a single session. If so, college students who are unable to commit to an 8-week program will still benefit tremendously from a toolbox of stress reduction techniques, especially during high-stress periods (e.g., finals).

The purpose of this study is to examine whether an acute bout of yoga, PMR, and DBE, delivered alone and in combination, are feasible and acceptable components in a single-session stress-reduction program for college students, and to explore initial effects on stress. We will use an efficient factorial design to gather data on the feasibility and acceptability of each of these three components, and to explore the initial main effects on stress.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate college students
* Aged 18 -24 years
* Capable of engaging in physical activity as assessed via the physical activity readiness questionnaire (PAR-Q+)
* Willing to provide consent and attend a single stress intervention session lasting up to 60 minutes
* Agree to all study procedures and assessments

Exclusion Criteria:

* Outside of 18-24 years of age
* Unable to safely engage in physical activity
* Not an undergraduate student at Wake Forest University
* Unwilling to complete study procedures

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Yield | Baseline
  Number consented/number contacted
Completion Rate | The day following the session
  Number completed/number consented
Acceptability of the intervention as assessed by survey | End of session
  Feedback survey of aspects of the program participants enjoyed and disliked

SECONDARY OUTCOMES:
Perceived acceptability of the intervention package as assessed by the Acceptability of Intervention Measure (AIM) | End of session
  A 4-item survey assessing perceived acceptability of a combination of intervention components
Perceived feasibility of delivering the intervention as assessed by the Feasibility of Intervention Measure (FIM) | End of session
  A 4-item survey assessing perceived feasibility of a combination of intervention components
Perceived appropriateness of the intervention package as assessed by the Intervention Appropriateness Measure (IAM) | End of session
  A 4-item survey assessing perceived appropriateness of a combination of intervention components
Perceived Stress | Pre-intervention, immediately preceding the single intervention session, immediately after completing the single intervention session, and 1 day after the single intervention session
  The Perceived Stress Scale: A 10-item scale assessing the participants' perceived stress with final scores falling between 0 and 40 such that higher scores reflect more stress.
Positive and negative affect | Pre-intervention, immediately preceding the single intervention session, immediately after completing the single intervention session, and 1 day after the single intervention session
  The Positive and Negative Affect Schedule (PANAS): An 20-item assessment of both positive and negative affect. The final scores are given on two subscales (positive affect and negative affect) ranging from 10-50 such that lower scores represent less of the affective state (i.e., less positive or negative affect) and 50 representing more of the affective state (i.e., more positive or negative affect).

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No